CLINICAL TRIAL: NCT04940416
Title: Oculometric Testing for the Diagnosis of Covert Hepatic Encephalopathy
Brief Title: Eye Movement Testing for Diagnosing Encephalopathy in Patients With Liver Disease
Status: Terminated | Type: Observational
Why Stopped: Collaboration between partners ended, covid
Sponsor: Stanford University (Other)
Collaborators: Neurofit Inc, Mountain View, California (Unknown)
Responsible Party: Principal Investigator, POkafor, Clinical Assistant Professor, Stanford University
Other Study IDs: 41796
Record Dates: First submitted 2021-06-17; First posted 2021-06-25 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Cirrhosis; Hepatic Encephalopathy
MeSH Terms: conditions — Fibrosis; Hepatic Encephalopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Cirrhosis: These will include patients with cirrhosis. They will perform the paper-based standard psychometric tests (number connection test A, number connection test B, line tracing test, and digital subtraction test, and serial dotting test, which take about 20 minutes). After completion of paper-based standard psychometric tests, participants will then perform the computer application test which takes about 5 minutes.
  Interventions: Device: Neurofit (oculometric testing)
- Non-cirrhosis: These will include patients without cirrhosis seen in the general gastroenterology clinic. Participants will perform the paper-based standard psychometric tests (number connection test A, number connection test B, line tracing test, and digital subtraction test, and serial dotting test, which take about 20 minutes). After completion of paper-based standard psychometric tests, participants will then perform the computer application test which takes about 5 minutes.
  Interventions: Device: Neurofit (oculometric testing)

INTERVENTIONS:
Device: Neurofit (oculometric testing) — The Neurofit test involves sitting on a chair with a head and chin rest to maintain stability. Patients will then follow a moving object on the computer screen with their eyes which allows estimation of individual oculometrics along with a composite score. No physical contact or placement of invasive devices will be performed. The total time for completion of all the tests is estimated at 30 minutes.

SUMMARY:
This study involves utilizing a noninvasive computer application (Neurofit) that performs oculometric assessment of dynamic visual processing in patients with liver cirrhosis to see if the presence of advance liver disease influences eye movement metrics.

DETAILED DESCRIPTION:
Cirrhosis is an increasingly prevalent medical condition in the United States that impacts health-related quality of life, healthcare resource utilization and survival. Patients with decompensated cirrhosis occasionally suffer from hepatic encephalopathy which is a serious complication that results from portosystemic shunting of blood leading to a spectrum of neuropsychiatric changes and alteration in consciousness levels when it becomes overt (overt hepatic encephalopathy, OHE).

Hepatic encephalopathy affects 30-45% of patients with cirrhosis and its occurrence and progression is associated with higher mortality.

In particular, Hepatic encephalopathy (HE) is an independent predictor of hospital readmissions in patients with cirrhosis. Encephalopathy could be overt with obvious deterioration in the level of consciousness leading to hospitalizations, but could also be covert and less obvious to the patient and healthcare provider.

Covert hepatic encephalopathy (CHE) is often unrecognized by healthcare providers leading to falls, motor vehicular accidents, and potential progression to overt confusion. Progression of CHE to OHE makes recognition of this condition important as early identification and treatment can potentially improve quality of life, reduce hospital readmissions and healthcare costs. Existing diagnostic tools are not only tedious and time consuming, but also impacted by factors such as level of education, reducing their utility in clinical practice. The ideal test would be easy to use, quantifiable, quick, cheap, reliable, and able to predict outcomes.

The exploratory study will utilize a noninvasive computer application (Neurofit) that performs oculometric assessment of dynamic visual processing. Eye movements are short latency, voluntary motor behaviors that consist of various aspects including visual motion, pursuit initiation, steady-state tracking, direction tuning, and speed tuning. The computer application is based on an eye movement methodology that can quantify many aspects of human dynamic visual processing using a noninvasive video-based eye tracking technology with validated oculometric analysis techniques.

Prior studies have demonstrated sensorimotor dysfunction in patients with diffuse brain injury which leads to derangement in information processing throughout the brain. This computer application has been utilized in patients with traumatic brain injury (TBI). Liston et al, in a study of 34 TBI patients, demonstrated that TBI patients had several individual oculometrics that were significantly deranged including pursuit latency, initial pursuit acceleration, pursuit gain, catch-up saccade amplitude, proportion smooth tracking, and speed responsiveness as compared to a separate control group. The application was able to discriminate TBI subjects from controls with an 81% probability that increased with self-reported TBI severity.

Rationale Hepatic encephalopathy is believed to occur as a consequence of portosystemic shunting leading to toxins, octapamines, free fatty acids amongst others accumulating in the brain, causing impairment in neurocognitive functioning. The extent of brain dysfunction associated with hepatic encephalopathy has not been fully characterized. Hepatic encephalopathy could potentially impair global brain function leading to oculomotor discoordination that can be detected with this computer software. By comparing individual and composite oculometric data between patients with cirrhosis and those without cirrhosis this study may identify any significant differences or distinct patterns that may exist as a result of hepatic encephalopathy. For this study, covert hepatic encephalopathy will be determined by paper-based psychometric testing. Any data obtained from this feasibility/exploratory study, will serve as preliminary data for larger studies and future validation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cirrhosis with clinical appointments in the pretransplant liver clinic
* Patients in the general gastroenterology clinic without a diagnosis of cirrhosis (controls)

Exclusion Criteria:

* Individuals <18 years
* cirrhotic patients with hepatocellular cancer
* individuals with uncontrolled neuropsychiatric illnesses or overt hepatic encephalopathy
* ongoing alcohol or illicit substance use
* non-English speakers, as the language barrier may impact psychometric test results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include consenting patients with cirrhosis seen in the gastroenterology and hematology clinic of the Stanford hospital. They will include patients with cirrhosis of varying severity. The non cirrhosis arm will include patients in the general gastroenterology clinic with no laboratory or radiological evidence of cirrhosis.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2021-06-17 (Actual); Study Completion 2021-06-17 (Actual)

PRIMARY OUTCOMES:
NeuroFit score | at first visit (up to 5 minutes)
  Composite oculometric test result

SECONDARY OUTCOMES:
Psychometric hepatic encephalopathy score | at first visit (up to 10 minutes)
  Composite score from paper based psychometric test

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University School of Medicine, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No